CLINICAL TRIAL: NCT02937805
Title: Effects of a Moisturizing Cream on Vaginal and Vulvar Mucous Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petra Larmo (Industry)
Collaborators: Turun Gynekologikeskus Oy (Unknown); Tekes - The Finnish Funding Agency for Technology and Innovation (Unknown)
Responsible Party: Sponsor-Investigator, Petra Larmo, R&D Manager, Aromtech Ltd.
Organization: Aromtech Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCMM
Record Dates: First submitted 2016-10-11; First posted 2016-10-19 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Vaginal Dryness; Vaginal Atrophy; Vulvar Dryness; Vulvar Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moisturizing vaginal and vulvar sea buckthorn oil cream (Experimental): Moisturizing non-hormonal vaginal and vulvar cream containing sea buckthorn oil as active ingredient (medical device product in development). Administered twice or once per day for 5 weeks. Post-menopausal women n= 55 + 45. Pre-menopausal women n=15
  Interventions: Device: Moisturizing vaginal and vulvar sea buckthorn oil cream
- Moisturizing vaginal and vulvar cream (Active Comparator): Moisturizing non-hormonal vaginal and vulvar cream (commercial medical device cream already on the market, not containing sea buckthorn oil). Administered once - twice per day for 5 weeks. Postmenopausal women n=55
  Interventions: Device: Moisturizing vaginal and vulvar cream
- Control (No Intervention): No moisturizing vaginal and vulvar cream for 5 weeks. Postmenopausal women n=55

INTERVENTIONS:
Device: Moisturizing vaginal and vulvar sea buckthorn oil cream
  Arms: Moisturizing vaginal and vulvar sea buckthorn oil cream
Device: Moisturizing vaginal and vulvar cream
  Arms: Moisturizing vaginal and vulvar cream

SUMMARY:
Vulvovaginal atrophy is a common problem associated with decreased levels of estrogen. Typical symptoms include feelings of dryness and uncomfort of the mucous membranes of intimate area. The objective of this study is to investigate the effects of a non-hormonal moisturizing cream on symptoms and signs of vulvovaginal atrophy and dryness.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of vaginal dryness, burning or itching
* Symptom severity at least moderate

Exclusion Criteria:

* Systemic hormonal replacement therapy during the last 12 months
* Local hormonal replacement therapy during the last 4 weeks
* Known allergy to ingredients of the study creams
* Pregnancy
* Breast-feeding

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of vaginal health index: scores of vaginal mucosa elasticity, fluid, pH, epithelial integrity, moisture | Baseline, 5 weeks
Change in vaginal and vulvar pH | Baseline, 5 weeks
Change in signs of vaginal and vulvar dryness: VAS evaluation by the study gynecologist | Baseline, 5 weeks
Change in signs of vaginal and vulvar mucosal integrity: VAS evaluation by the study gynecologist | Baseline, 5 weeks
Change in signs of vaginal and vulvar inflammation and irritation: VAS evaluation by the study gynecologist | Baseline, 5 weeks
Change in symptoms of vaginal and vulvar atrophy and dryness: symptom questionnaires; scoring from 0 to 3 dryness, burning, itching; VAS evaluation of mucosal dryness, irritation, soreness, pain during exercise, pain during intercourse | Baseline, 5 weeks

SECONDARY OUTCOMES:
Change in symptoms of vaginal and vulvar atrophy and dryness: symptom logbooks; daily scoring from 0 to 3 dryness, burning, itching, pain, soreness, symptoms during intercourse | From baseline to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Risto Erkkola, Professor, Principal Investigator — Turun Gynekologikeskus
Locations (1):
- Turun Gynekologikeskus, Turku, Finland

IPD SHARING:
Plan to Share IPD: No